CLINICAL TRIAL: NCT05256381
Title: A Phase 2, Open-label, Single-arm, Multicenter Study of SOT101 in Combination With Pembrolizumab to Evaluate the Efficacy and Safety in Patients With Selected Advanced/Refractory Solid Tumors
Brief Title: A Study of SOT101 in Combination With Pembrolizumab to Evaluate the Efficacy and Safety in Patients With Selected Advanced Solid Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to lack of expected efficacy shown at the time of the interim analysis
Sponsor: SOTIO Biotech AG (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Sotio Biotech Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC104; KEYNOTE-D13 (Other: Merck Sharp & Dohme); AURELIO-04 (Other: SOTIO Biotech AG); 2021-005774-25 (EudraCT Number); MK-3475-D13 (Other: Merck Sharp & Dohme)
Record Dates: First submitted 2022-02-08; First posted 2022-02-25 (Actual); Results first posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer; Colorectal Cancer; Cutaneous Squamous Cell Carcinoma; Hepatocellular Carcinoma; Castration-resistant Prostate Cancer; Ovarian Cancer
Keywords: SOT101; SO-C101; Pembrolizumab; Non-Small Cell Lung Cancer; Colorectal Cancer; Cutaneous Squamous Cell Carcinoma; Advanced Hepatocellular Carcinoma; Metastatic Castration-resistant Prostate Cancer; Ovarian Cancer; KEYNOTE-D13; AURELIO-04; Nanrilkefusp Alfa
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Carcinoma, Hepatocellular; Ovarian Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nanrilkefusp Alfa and Pembrolizumab (Experimental): Participants will be treated with 12 μg/kg of nanrilkefusp alfa on Day 1, Day 2, Day 8, and Day 9 of each 3-week cycle in combination with 200 mg pembrolizumab on Day 1 of each 3-week cycle.
  Interventions: Drug: Nanrilkefusp Alfa; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Nanrilkefusp Alfa — Subcutaneous (SC) injection.
  Other Names: SOT101
Drug: Pembrolizumab — Intravenous (IV) infusion via peripheral or central venous line.
  Other Names: KEYTRUDA®

SUMMARY:
The primary objective of the study is to estimate the antitumor efficacy of nanrilkefusp alfa in combination with pembrolizumab in selected tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participants with the following histologically or cytologically confirmed solid tumor indications and line of treatment:

  1. Non-small cell lung cancer (NSCLC).
  2. Colorectal cancer.
  3. Cutaneous squamous cell carcinoma (cSCC).
  4. Advanced hepatocellular carcinoma (not applicable in France).
  5. mCRPC.
  6. Ovarian cancer.
* Have measurable disease per RECIST 1.1. mCRPC participants with no measurable disease and only widespread bone disease must have a CTC count of ≥5 cells per 7.5 mL of blood.
* Availability of tumor tissue from a fresh biopsy at screening unless the biopsy cannot be obtained due to safety reasons or non-accessibility of the tumor site. If it is not possible to obtain a fresh biopsy, every effort should be taken to retrieve an archival biopsy. Archived, fixed tumor tissue may only be collected if taken preferentially after completion of the most recent systemic tumor therapy and within 12 months prior to the first dose of study treatment.
* Eastern Cooperative Oncology Group (ECOG) score 0-1.
* Have recovered from all AEs (except alopecia) due to previous therapies to grade ≤1 (excluding alopecia) or have stable grade 2 neuropathy.
* Have adequate organ function as defined below:

  1. Hematology:

     1. Absolute neutrophil count ≥1500/μL.
     2. Platelets ≥100 000/μL.
     3. Hemoglobin ≥9.0 g/dL .
  2. Renal function: Creatinine clearance as measured by glomerular filtration rate ≥30 mL/min using Cockcroft-Gault equation.
  3. Hepatic function: Alanine transaminase (ALT)/aspartate transaminase (AST) ≤2.5× upper limit of normal (ULN) and total bilirubin ≤1.5×ULN or direct bilirubin ≤ ULN in participants without liver metastasis. In participants with liver metastasis, ALT/AST ≤5×ULN is allowed but total bilirubin must be ≤2×ULN.
  4. Prothrombin time and activated partial thromboplastin time ≤1.5×ULN.
* Participants must not have active hepatitis B or hepatitis C infection.
* Adequate contraception must be applied in all women of childbearing potential (WOCBP) and in male participants.

Exclusion Criteria:

* Has received prior therapy with an anti-programmed cell death protein 1 (anti-PD-1), anti-programmed cell death ligand 1 (anti-PD-L1), or anti-programmed cell death ligand 2 (anti-PD-L2) agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor and was discontinued from that treatment due to a grade ≥3 AE.
* Prior exposure to agonists of interleukin (IL)-2 or IL-15.
* Prior systemic anti-cancer therapies, including investigational agents:

  1. Less than 4 weeks for systemic chemotherapy and immuno-oncology therapies; and for tyrosine kinase inhibitors 4 weeks or 5 half-lives (whichever is shorter).
  2. Less than 4 weeks from major surgeries and not recovered adequately.
* Has received prior radiotherapy within 2 weeks of the start of study interventions or have had a history of radiation pneumonitis.
* NSCLC indication only: Received radiation therapy to the lung >30 Gy within 6 months.
* Has received a live or live-attenuated vaccine within 30 days.
* Clinically significant cardiac abnormalities including prior history of any of the following:

  1. Cardiomyopathy, with left ventricular ejection fraction ≤ 50%.
  2. Congestive heart failure of New York Heart Association grade ≥2.
  3. History of clinically significant artery or coronary heart disease.
  4. Prolongation of QTcF >450 msec .
  5. Clinically significant cardiac arrythmia that cannot be controlled with adequate medication.
* Uncontrolled hypertension defined as systolic blood pressure >160 mmHg, diastolic blood pressure >110 mmHg.
* Prior allogeneic hematopoietic stem cell transplantation within the last 5 years.
* Prior allogeneic tissue/solid organ transplant.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy.
* History of or serology positive for human immunodeficiency virus (HIV).
* Has a known additional malignancy that is progressing or has required active treatment within the past 5 years, except for basal cell carcinoma of the skin or carcinoma in situ that have undergone potentially curative therapy are not excluded.
* Has known active central nervous system metastases and/or carcinomatous meningitis, unless stable.
* Had severe hypersensitivity (grade ≥3) to pembrolizumab and/or any of its excipients.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years.
* History of (non-infectious) pneumonitis/interstitial lung disease that required steroids or current pneumonitis/interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has any condition that might confound the results of the study or interfere with the participant's participation for the full duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-11-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (54):
- United States (2):
  - Innovative Clinical Research Institute, Whittier, California
  - University of Pittsburg Medical Center (UPMC) Hillman Cancer Center, Pittsburgh, Pennsylvania
- Belgium (5):
  - Institut Jules Bordet, Anderlecht
  - Cliniques Universitaires Saint-Luc, Brussels
  - Grand Hospital de Charleroi, Charleroi
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
- Czechia (3):
  - Masarykuv Onkologicky Ustav, Brno
  - Nemocnice Hořovice, Hořovice
  - Fakultní nemocnice Olomouc, Olomouc
- France (12):
  - Hôpital Ambroise-Paré, Boulogne-Billancourt
  - Merchant Logo Institute Bergonié, Bourdeaux
  - Centre de Lutte Contre le Cancer, Caen
  - Centre Francois Baclesser, Caen
  - Hospital del la Timone, Marseille
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Centre Antoine Lacassagne, Nice
  - Hospital L'archet, Nice
  - Hôpital Foch, Suresnes
  - Institut Universitaire du Cancer de Toulouse Oncopole, Toulouse
  - Institute Claudius Regaud, Toulouse
  - Gustave Roussy, Villejuif
- Georgia (9):
  - High Technology Hospital MedCenter Ltd - Batumi, Batumi
  - Evex Hospitals- Kutaisi Referral, Kutaisi
  - LLC Todua Clinic, Tbilisi
  - Evex Hospitals - Caraps Medline, Tbilisi
  - New Vision University Hospital, Tbilisi
  - Tbilisi Institute of Medicine, Tbilisi
  - Jerarsi Clinic, Tbilisi
  - Consilium Medulla Multiprofile Clinic, Tbilisi
  - Evex Hospitals - Caucasus Medical Center, Tbilisi
- Hungary (2):
  - Észak-Pesti Centrumkórház - Honvédkórház, Budapest
  - Petz Aladár Egyetemi Oktató Kórház - Győr, Győr
- Italy (8):
  - Azienda Socio Sanitaria Territoriale (ASST) degli Spedali Civili di Brescia, Brescia
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST, Meldola
  - Instituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli
  - Ospedale Guglielmo da Saliceto, Piacenza
  - Fondazione Policlinico Universitario Agostino Gemelli, Rome
  - Azienda Ospedaliera Universitaria Senese - L'ospedale Santa Maria alle Scotte, Siena
  - Ospedale Civile di Sondrio, Sondrio
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Poland (3):
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan, Greater Poland Voivodeship
  - Pratia Poznań, Skorzewo
  - MTZ Clinical Research powered by Pratia, Warsaw
- Spain (10):
  - Hospital Teresa Herrera - Materno Infantil, A Coruña
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Institut Catala d'Oncologia, Barcelona
  - Clinica Universidad de Navarra - Pamplona, Madrid
  - Clínica Universidad de Navarra - Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Madrid
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-small Cell Lung Cancer: Advanced and/or metastatic non-small cell lung cancer with disease progression on or after an immune checkpoint inhibitor-containing regimen and a platinum-containing regimen, with no epidermal growth factor receptor or anaplastic lymphoma kinase genomic tumor aberrations, and who were not amenable to curative treatment
- Colorectal Cancer: Microsatellite instability-high or mismatch repair deficient colorectal cancer that was unresectable or metastatic
- Cutaneous Squamous Cell Carcinoma: Recurrent or metastatic cutaneous squamous cell carcinoma that was not curable by surgery or radiation and in second line if refractory or relapsed after a checkpoint inhibitor-containing regimen and radiotherapy was not feasible
- Hepatocellular Carcinoma: Advanced hepatocellular carcinoma after recurrence or failure of an immune checkpoint inhibitor (not applicable in France)
- Metastatic Castration-resistant Prostate Cancer: Treatment-refractory metastatic castration-resistant prostate cancer after recurrence or failure of docetaxel and prior treatment with abiraterone, enzalutamide, or any other androgen receptor-targeted agent
- Ovarian Cancer: Advanced recurrent ovarian cancer after recurrence or failure on the last platinum-based therapy within 6 months
Period: Overall Study
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer
Started | 40 | 8 | 12 | 12 | 55 | 39
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 40 | 8 | 12 | 12 | 55 | 39
Not completed — Withdrawal by Subject | 4 | 0 | 2 | 2 | 8 | 6
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 2 | 0
Not completed — Death | 17 | 3 | 4 | 5 | 24 | 21
Not completed — Other, not specified | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Study terminated by sponsor | 18 | 5 | 5 | 5 | 18 | 11
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: 1 patient in the Metastatic castration-resistant prostate cancer withdrew from the trial before any baseline and other data could be collected. This patient did not start any treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer | Total
Number analyzed (Participants) | 40 | 8 | 12 | 12 | 54 | 39 | 165
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 5 | 1 | 8 | 14 | 21 | 72
  >=65 years | 17 | 3 | 11 | 4 | 40 | 18 | 93
Age, Continuous [Median (Standard Deviation); unit: years] | 63.5 (10.43) | 59.0 (18.34) | 75.5 (10.95) | 63.5 (11.02) | 68.0 (6.57) | 64.0 (11.59) | 66.0 (10.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 3 | 2 | 1 | 0 | 39 | 57
  Male | 28 | 5 | 10 | 11 | 54 | 0 | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 0 | 1 | 0 | 4
  Not Hispanic or Latino | 30 | 6 | 9 | 12 | 48 | 35 | 140
  Unknown or Not Reported | 8 | 1 | 3 | 0 | 5 | 4 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 32 | 7 | 9 | 12 | 49 | 36 | 145
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 8 | 1 | 3 | 0 | 4 | 3 | 19
Region of Enrollment [Number; unit: participants]
  Belgium | 6 | 0 | 0 | 4 | 1 | 8 | 19
  Hungary | 0 | 0 | 0 | 0 | 2 | 0 | 2
  United States | 1 | 0 | 0 | 0 | 2 | 1 | 4
  Czechia | 2 | 1 | 0 | 0 | 2 | 3 | 8
  Poland | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Italy | 4 | 0 | 2 | 0 | 2 | 0 | 8
  Georgia | 13 | 4 | 6 | 8 | 19 | 6 | 56
  France | 8 | 1 | 3 | 0 | 4 | 5 | 21
  Spain | 6 | 1 | 1 | 0 | 21 | 16 | 45

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Objective Response Rate According to Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1)
Time Frame: Day 1 up to approximately 2 years and 2 months
Population: All patients exposed to the combination therapy for at least one treatment cycle. This is defined as patients with 4 doses of SOT101 and 1 dose of pembrolizumab in Cycle 1, or patients exposed to both SOT101 and pembrolizumab in Cycle 1 who started Cycle 2. Only patients with measurable disease at baseline were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer
Number analyzed (Participants) | 39 | 6 | 11 | 11 | 40 | 35
percentage of participants | 5.1 [0.6 to 17.3] | 33.3 [4.3 to 77.7] | 27.3 [6.0 to 61.0] | 0 [0 to 28.5] | 10.0 [2.8 to 23.7] | 11.4 [3.2 to 26.7]

2. Secondary Outcome: Number of Patients With a Treatment-emergent Adverse Event
Time Frame: Day 1 up to approximately 2 years and 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer
Number analyzed (Participants) | 40 | 8 | 12 | 12 | 54 | 39
Participants | 40 | 8 | 12 | 12 | 54 | 39

3. Secondary Outcome: Number of Patients With an Adverse Event of Special Interest
Time Frame: Day 1 up to approximately 2 years and 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer
Number analyzed (Participants) | 40 | 8 | 12 | 12 | 54 | 39
Participants | 0 | 1 | 0 | 0 | 0 | 0

4. Secondary Outcome: Percentage of Patients With Objective Response Rate According to RECIST for Immune-based Therapeutics (iRECIST)
Time Frame: Day 1 up to approximately 2 years and 2 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer
Number analyzed (Participants) | 39 | 6 | 11 | 11 | 40 | 35
percentage of participants | 7.7 [1.6 to 20.9] | 33.3 [4.3 to 77.7] | 36.4 [10.9 to 69.2] | 0 [0 to 28.5] | 12.5 [4.2 to 26.8] | 11.4 [3.2 to 26.7]

5. Secondary Outcome: Number of Patients With Best Overall Response According to RECIST 1.1: Complete Response
Time Frame: Day 1 up to approximately 2 years and 2 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer
Number analyzed (Participants) | 39 | 6 | 11 | 11 | 40 | 35
Participants | 0 | 0 | 1 | 0 | 0 | 0

6. Secondary Outcome: Number of Patients With Best Overall Response According to RECIST 1.1: Partial Response
Time Frame: Day 1 up to approximately 2 years and 2 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer
Number analyzed (Participants) | 39 | 6 | 11 | 11 | 40 | 35
Participants | 2 | 2 | 2 | 0 | 4 | 4

7. Secondary Outcome: Number of Patients With Best Overall Response According to RECIST 1.1: Stable Disease
Time Frame: Day 1 up to approximately 2 years and 2 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer
Number analyzed (Participants) | 39 | 6 | 11 | 11 | 40 | 35
Participants | 12 | 3 | 2 | 5 | 14 | 4

8. Secondary Outcome: Number of Patients With Best Overall Response According to RECIST 1.1: Progressive Disease
Time Frame: Day 1 up to approximately 2 years and 2 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer
Number analyzed (Participants) | 39 | 6 | 11 | 11 | 40 | 35
Participants | 20 | 1 | 6 | 5 | 18 | 23

9. Secondary Outcome: Number of Patients With Best Overall Response According to iRECIST: Complete Response
Time Frame: Day 1 up to approximately 2 years and 2 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer
Number analyzed (Participants) | 39 | 6 | 11 | 11 | 40 | 35
Participants | 0 | 0 | 1 | 0 | 0 | 0

10. Secondary Outcome: Number of Patients With Best Overall Response According to iRECIST: Partial Response
Time Frame: Day 1 up to approximately 2 years and 2 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer
Number analyzed (Participants) | 39 | 6 | 11 | 11 | 40 | 35
Participants | 3 | 2 | 3 | 0 | 5 | 4

11. Secondary Outcome: Number of Patients With Best Overall Response According to iRECIST: Stable Disease
Time Frame: Day 1 up to approximately 2 years and 2 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer
Number analyzed (Participants) | 39 | 6 | 11 | 11 | 40 | 35
Participants | 15 | 3 | 2 | 5 | 15 | 4

12. Secondary Outcome: Number of Patients With Best Overall Response According to iRECIST: Unconfirmed Progressive Disease
Time Frame: Day 1 up to approximately 2 years and 2 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer
Number analyzed (Participants) | 39 | 6 | 11 | 11 | 40 | 35
Participants | 13 | 0 | 3 | 4 | 14 | 15

13. Secondary Outcome: Number of Patients With Best Overall Response According to iRECIST: Confirmed Progressive Disease
Time Frame: Day 1 up to approximately 2 years and 2 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer
Number analyzed (Participants) | 39 | 6 | 11 | 11 | 40 | 35
Participants | 3 | 1 | 2 | 1 | 2 | 8

14. Secondary Outcome: Duration of Response According to RECIST 1.1
Time Frame: Day 1 up to approximately 2 years and 2 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer
Number analyzed (Participants) | 39 | 6 | 11 | 11 | 40 | 35
months | 3.6 [1.7 to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [2.8 to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [4.3 to NA] — Insufficient number of participants with events | 3.0 [2.8 to NA] — Insufficient number of participants with events

15. Secondary Outcome: Duration of Response According to iRECIST
Time Frame: Day 1 up to approximately 2 years and 2 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer
Number analyzed (Participants) | 39 | 6 | 11 | 11 | 40 | 35
months | 3.6 [1.7 to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [2.8 to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | 13.9 [4.3 to NA] — Insufficient number of participants with events | 3.0 [2.8 to NA] — Insufficient number of participants with events

16. Secondary Outcome: Percentage of Patients With Clinical Benefit Rate According to RECIST 1.1
Time Frame: Day 1 up to approximately 2 years and 2 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer
Number analyzed (Participants) | 39 | 6 | 11 | 11 | 40 | 35
percentage of participants | 35.9 [21.2 to 52.8] | 83.3 [35.9 to 99.6] | 45.5 [16.7 to 76.6] | 45.5 [16.7 to 76.6] | 45.0 [29.3 to 61.5] | 22.9 [10.4 to 40.1]

17. Secondary Outcome: Percentage of Patients With Clinical Benefit Rate According to iRECIST
Time Frame: Day 1 up to approximately 2 years and 2 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer
Number analyzed (Participants) | 39 | 6 | 11 | 11 | 40 | 35
percentage of participants | 46.2 [30.1 to 62.8] | 83.3 [35.9 to 99.6] | 54.5 [23.4 to 83.3] | 45.5 [16.7 to 76.6] | 50.0 [33.8 to 66.2] | 22.9 [10.4 to 40.1]

18. Secondary Outcome: Progression-free Survival According to RECIST 1.1
Time Frame: Day 1 up to approximately 2 years and 2 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer
Number analyzed (Participants) | 39 | 6 | 11 | 11 | 40 | 35
months | 1.6 [1.3 to 2.8] | NA [1.1 to NA] — Insufficient number of participants with events | 1.4 [1.2 to NA] — Insufficient number of participants with events | 2.7 [1.1 to 4.3] | 2.6 [1.4 to 6.4] | 1.6 [1.4 to 2.6]

19. Secondary Outcome: Progression-free Survival According to iRECIST
Time Frame: Day 1 up to approximately 2 years and 2 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer
Number analyzed (Participants) | 39 | 6 | 11 | 11 | 40 | 35
months | 3.0 [1.3 to 5.7] | NA [1.1 to NA] — Insufficient number of participants with events | 4.1 [1.2 to NA] — Insufficient number of participants with events | 2.7 [1.1 to 4.3] | 4.6 [1.6 to 6.8] | 1.6 [1.4 to 2.6]

20. Secondary Outcome: Time to Response According to RECIST 1.1
Time Frame: Day 1 up to approximately 2 years and 2 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer
Number analyzed (Participants) | 39 | 6 | 11 | 11 | 40 | 35
months | NA [NA to NA] — Insufficient number of participants with events | 14.1 [1.6 to NA] — Insufficient number of participants with events | NA [1.4 to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [6.9 to NA] — Insufficient number of participants with events

21. Secondary Outcome: Time to Response According to iRECIST
Time Frame: Day 1 up to approximately 2 years and 2 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer
Number analyzed (Participants) | 39 | 6 | 11 | 11 | 40 | 35
months | NA [NA to NA] — Insufficient number of participants with events | 14.1 [1.6 to NA] — Insufficient number of participants with events | NA [1.4 to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [6.9 to NA] — Insufficient number of participants with events

22. Secondary Outcome: Duration of Response According to Prostate Cancer Clinical Trials Working Group 3 Modified RECIST 1.1
Time Frame: Day 1 up to approximately 2 years and 2 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Metastatic Castration-resistant Prostate Cancer
Number analyzed (Participants) | 40
months | NA [4.3 to NA] — Insufficient number of participants with events

23. Secondary Outcome: Percentage of Patients With Clinical Benefit Rate According to Prostate Cancer Clinical Trials Working Group 3 Modified RECIST 1.1
Time Frame: Day 1 up to approximately 2 years and 2 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Metastatic Castration-resistant Prostate Cancer
Number analyzed (Participants) | 40
percentage of participants | 45.0 [29.3 to 61.5]

24. Secondary Outcome: Progression-free Survival According to Prostate Cancer Clinical Trials Working Group 3 Modified RECIST 1.1
Time Frame: Day 1 up to approximately 2 years and 2 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Metastatic Castration-resistant Prostate Cancer
Number analyzed (Participants) | 40
months | 2.6 [1.4 to 6.4]

25. Secondary Outcome: Percentage of Patients With Circulating Tumor Cell Count Conversion as Assessed According to Prostate Cancer Clinical Trials Working Group 3 Modified RECIST 1.1
Time Frame: Day 1 up to approximately 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Metastatic Castration-resistant Prostate Cancer
Number analyzed (Participants) | 40
percentage of participants | 3.8 [0.5 to 13.2]

26. Secondary Outcome: Percentage of Patients With Confirmed Prostate-specific Antigen Decline of ≥50% as Assessed According to Prostate Cancer Clinical Trials Working Group 3 Modified RECIST 1.1
Time Frame: Day 1 up to approximately 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Metastatic Castration-resistant Prostate Cancer
Number analyzed (Participants) | 40
percentage of participants | 13.5 [5.8 to 26.7]

27. Secondary Outcome: Time to Confirmed Prostate-specific Antigen Progression as Assessed According to Prostate Cancer Clinical Trials Working Group 3 Modified RECIST 1.1
Time Frame: Day 1 up to approximately 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Metastatic Castration-resistant Prostate Cancer
Number analyzed (Participants) | 40
months | 2.3 [1.3 to 4.3]

28. Secondary Outcome: Nanrilkefusp Alfa Concentration Profile, Cycle 1 Day 1, 30 (+/-5) Minutes After Nanrilkefusp Alfa Administration
Time Frame: Cycle 1 Day 1, 30 (+/-5) minutes after nanrilkefusp alfa administration
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer
Number analyzed (Participants) | 37 | 8 | 12 | 12 | 53 | 38
ng/mL | 1.0900 [0.260 to 3.850] | 0.5890 [0.487 to 4.530] | 0.7200 [0.363 to 5.580] | 0.9470 [0.358 to 3.460] | 0 [0 to 4.370] | 0.9020 [0.151 to 3.690]

29. Secondary Outcome: Nanrilkefusp Alfa Concentration Profile, Cycle 1 Day 1, 2 Hours (+/-15 Minutes) After Nanrilkefusp Alfa Administration
Time Frame: Cycle 1 Day 1, 2 hours (+/-15 minutes) after nanrilkefusp alfa administration
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer
Number analyzed (Participants) | 37 | 8 | 12 | 12 | 53 | 38
ng/mL | 3.6800 [0.628 to 15.600] | 3.6700 [1.220 to 11.900] | 3.4250 [1.350 to 19.100] | 2.5600 [0.820 to 4.070] | 3.4500 [0.291 to 15.800] | 3.1300 [0.288 to 10.700]

30. Secondary Outcome: Number of Patients With Anti-drug Antibodies, Cycle 4 Day 1
Time Frame: Cycle 4 Day 1, approximately 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer
Number analyzed (Participants) | 39 | 8 | 12 | 12 | 53 | 39
Participants | 5 | 3 | 3 | 0 | 4 | 5

ADVERSE EVENTS:
Time Frame: Day 1 up to approximately 2 years and 2 months
Description: Only treatment-emergent AEs (TEAEs) were analyzed (see the definition above); the tables include information on TEAEs, serious TEAEs, and all deaths; causality was assessed by investigators. All-cause mortality was assessed in Enrolled patients (all who signed the ICF) whereas AEs were assessed in All-subjects-as-treated (all who were treated with nanrilkefusp alfa or pembrolizumab).
Arm/Group | Non-small Cell Lung Cancer | Colorectal Cancer | Cutaneous Squamous Cell Carcinoma | Hepatocellular Carcinoma | Metastatic Castration-resistant Prostate Cancer | Ovarian Cancer
All-Cause Mortality (participants affected / at risk) | 17/40 | 3/8 | 4/12 | 5/12 | 24/55 | 21/39
Serious Adverse Events (participants affected / at risk) | 23/40 | 3/8 | 3/12 | 3/12 | 28/54 | 28/39
Other Adverse Events (participants affected / at risk) | 40/40 | 8/8 | 12/12 | 12/12 | 54/54 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-small Cell Lung Cancer (N=40) | Colorectal Cancer (N=8) | Cutaneous Squamous Cell Carcinoma (N=12) | Hepatocellular Carcinoma (N=12) | Metastatic Castration-resistant Prostate Cancer (N=54) | Ovarian Cancer (N=39)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 7 (7) | 6 (6)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 8 (14)
General physical health deterioration (General disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — 2 SAEs were classified by the investigator as Unknown cause of death. Both were coded per MedDRA as General disorders and administration site conditions/Death.
Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 2 (6) | 1 (1) | 3 (4) | 1 (3) | 7 (9) | 7 (7)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-small Cell Lung Cancer (N=40) | Colorectal Cancer (N=8) | Cutaneous Squamous Cell Carcinoma (N=12) | Hepatocellular Carcinoma (N=12) | Metastatic Castration-resistant Prostate Cancer (N=54) | Ovarian Cancer (N=39)
Lymphocyte count decreased (Investigations) | 17 (26) | 5 (10) | 4 (10) | 8 (14) | 21 (42) | 7 (9)
Aspartate aminotransferase increased (Investigations) | 15 (23) | 3 (4) | 1 (1) | 1 (5) | 16 (30) | 9 (10)
Alanine aminotransferase increased (Investigations) | 14 (22) | 2 (3) | 1 (1) | 2 (2) | 14 (17) | 9 (11)
Blood bilirubin increased (Investigations) | 5 (6) | 1 (3) | 0 (0) | 3 (4) | 8 (9) | 3 (5)
Neutrophil count decreased (Investigations) | 1 (3) | 2 (7) | 2 (5) | 2 (3) | 10 (24) | 3 (10)
Platelet count decreased (Investigations) | 3 (4) | 0 (0) | 0 (0) | 3 (6) | 11 (32) | 1 (1)
Blood creatinine increased (Investigations) | 4 (5) | 1 (2) | 2 (2) | 1 (4) | 6 (17) | 2 (6)
Blood alkaline phosphatase increased (Investigations) | 8 (11) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Amylase increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (13) | 4 (4)
Weight decreased (Investigations) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Lipase increased (Investigations) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Hypotension (Vascular disorders) | 9 (11) | 2 (4) | 2 (7) | 0 (0) | 14 (43) | 5 (5)
Hypertension (Vascular disorders) | 4 (4) | 0 (0) | 2 (2) | 3 (4) | 3 (4) | 4 (4)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 4 (4)
Headache (Nervous system disorders) | 6 (6) | 1 (3) | 1 (5) | 0 (0) | 5 (8) | 5 (8)
Tremor (Nervous system disorders) | 4 (5) | 1 (1) | 0 (0) | 1 (1) | 8 (14) | 2 (3)
Pyrexia (General disorders) | 26 (114) | 4 (40) | 10 (30) | 7 (19) | 38 (161) | 36 (154)
Chills (General disorders) | 15 (20) | 3 (12) | 3 (11) | 1 (1) | 21 (32) | 15 (54)
Fatigue (General disorders) | 15 (16) | 1 (1) | 3 (4) | 6 (6) | 13 (20) | 14 (18)
Injection site reaction (General disorders) | 11 (48) | 3 (9) | 2 (3) | 4 (7) | 13 (25) | 19 (92)
Asthenia (General disorders) | 12 (12) | 1 (1) | 4 (6) | 1 (2) | 20 (25) | 13 (17)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 4 (4)
Chest pain (General disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 17 (23) | 1 (1) | 1 (3) | 3 (4) | 31 (52) | 8 (9)
Cytokine release syndrome (Immune system disorders) | 6 (23) | 2 (10) | 2 (4) | 1 (3) | 12 (38) | 2 (7)
Vomiting (Gastrointestinal disorders) | 11 (14) | 0 (0) | 1 (1) | 4 (7) | 17 (33) | 22 (43)
Nausea (Gastrointestinal disorders) | 10 (18) | 1 (19) | 2 (2) | 2 (5) | 13 (20) | 24 (36)
Diarrhoea (Gastrointestinal disorders) | 5 (8) | 1 (8) | 1 (1) | 3 (3) | 4 (5) | 12 (15)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 7 (8)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 10 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 6 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 3 (3)
Hypothyroidism (Endocrine disorders) | 3 (4) | 1 (1) | 1 (1) | 1 (2) | 6 (6) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (3) | 1 (3) | 2 (2) | 4 (6) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (6) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 11 (12) | 0 (0) | 1 (1) | 2 (2) | 11 (13) | 10 (11)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 0 (0) | 2 (3) | 6 (9) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 12 (19) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (7) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (11) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this clinical trial will be published and/or presented at scientific meetings in their totality in a timely manner. Any formal publication of clinical trial results will be a collaborative effort between the sponsor and the investigator(s). All manuscripts or abstracts will be reviewed and approved in written by the sponsor before submission. The sponsor may request a delay in publication if there are important intellectual property concerns.

DOCUMENTS (2):
  • Study Protocol (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT05256381/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT05256381/SAP_001.pdf